CLINICAL TRIAL: NCT07262060
Title: Optimizing Caffeine Therapy for Hypoxia in Preterm Neonates: A Randomized Trial Assessing Efficacy, Acute Kidney and Brain Injury, Safety, and Pharmacokinetics
Brief Title: Improving Preterm Kidney Outcomes With Caffeine
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-1079; Protocol Version 10/9/2025 (Other: UW Madison); SMPH\PEDIATRICS\NEONATO (Other: UW Madison); 1R01HD116793-01 (NIH)
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Kidney Injury; Pre-Term
Keywords: caffeine; acute kidney injury
MeSH Terms: conditions — Premature Birth; Acute Kidney Injury | interventions — caffeine citrate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, double blind, single-center trial of the effectiveness of additional caffeine compared to placebo in preterm neonates less than 30 weeks gestational age.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Caffeine (Experimental)
  Interventions: Drug: Caffeine citrate
- Arm 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 3: Control (No Intervention)

INTERVENTIONS:
Drug: Caffeine citrate — intravenous (IV) caffeine citrate (20 milligrams per kilogram) (n = 45) followed by 8 milligrams per kilogram daily maintenance
  Arms: Arm 1: Caffeine
Drug: Placebo — same volume of 0.9 percent Sodium Chloride United States Pharmacopeia (USP) (n=45)
  Other Names: saline
  Arms: Arm 2: Placebo

SUMMARY:
This study is being done to see if additional caffeine citrate (20 milligrams per kilogram IV bolus) helps babies with low kidney oxygenation already being treated with caffeine citrate (20 milligrams per kilogram IV bolus on day of life (DOL) 1 followed by 8 milligrams per kilogram daily maintenance). The investigators hypothesize that additional caffeine will improve kidney oxygen levels, while not causing any brain injury, and may reduce rates of acute kidney injury compared to placebo. This study will take place in preterm babies born less than 30 weeks gestational age, with the intervention occurring between greater than 48 hours of age until DOL 14 and outcomes tracked until neonatal intensive care unit (NICU) discharge.

DETAILED DESCRIPTION:
The study population will consist of 102 preterm neonates born less than 30 weeks gestational age who have an intravenous (IV) line for which IV medications can be administered and who can have brain and kidney Near Infrared Spectroscopy (NIRS) monitoring.

Eligible participants will be enrolled between 12-96 hours of life after preterm birth and admission to the Meriter NICU. Baseline data will be collected and NIRS monitoring will be started when appropriate as determined by the team based on clinical guidelines and standard of care.

Those participants having kidney oxygenation less than 50 percent (and troubleshooting procedures have occurred and while ensuring brain oxygenation is not below 55 percent) after 48 hours and within the first 14 DOL will be randomized in a 1:1 manner to one of two treatment arms (Arm 1 and Arm 2).

* Arm 1: IV caffeine citrate (20 mg/kg) (n = 45)
* Arm 2: Placebo - same volume of 0.9% Sodium Chloride United States Pharmacopeia (USP) (n=45)

Those participants who do not develop kidney hypoxia during the first 14 DOL will be the normal kidney oxygenation control group and receive no intervention (Arm 3).

* Arm 3: Normal Kidney oxygenation (no intervention) (Approximately n = 12)

Participant accrual will occur over 48 months. Participants will complete all study specific activities during the NICU hospitalization over the course of the first 28 DOL and clinical outcomes will be collected through NICU discharge or 6 months of age, whichever occurs first. Each participant will contribute blood specimens for creatinine and caffeine levels as well as approximately 20-40 urine samples for biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth between 23 0/7 and 29 6/7 weeks.
* Able to have near-infrared spectroscopy (NIRS) monitoring of cerebral and kidney oxygenation.
* Able to receive IV medications.
* Indwelling umbilical arterial catheter (UAC), umbilical venous catheter (UVC), peripheral arterial line (PAL), or peripherally inserted central catheter (PICC) already in place that can draw blood.
* Receiving caffeine at the time of enrollment
* Have a birth parent who is at least 18 years old and have a parent or guardian who is able to provide parental permission in English or Spanish

Exclusion Criteria:

* Known or suspected major congenital anomaly of the brain, heart, lungs or kidney (excluding UTD A1 pyelectasis).
* Known or suspected chromosomal or genetic anomaly.
* Not suitable for study participation due to other reasons at the discretion of the investigators.

Ages: 12 Hours to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Improvement in Kidney Oxygenation | Up to 3 hours post-intervention (Between days 1 and 17)
  In the 3 hours after receiving the intervention or placebo, participants have kidney oxygenation monitored. Improvement in oxygenation is defined as having 30 minutes where at least 90 percent of measured values are at least 50 percent.

SECONDARY OUTCOMES:
Number of Days of Acute Kidney Injury (AKI) | 14 days after intervention
  AKI as defined by the Kidney Disease Improving Global Outcomes (KDIGO) foundation. Outcome is measured for the 14 days after intervention.
Proportion of Participants with a Sustained Decrease in Cerebral Oxygenation | up to 3 hours post-intervention (Between days 1 and 17)
  In the 3 hours after receiving the intervention or placebo, participants have cerebral oxygenation monitored. A sustained decrease in cerebral oxygenation is defined as less than 60 percent oxygenation for at least 60 minutes.

OTHER OUTCOMES:
Change in Urinary Biomarker Concentrations | baseline, day 17
Rates of Brain Injury | up to 6 months
  Rates of Brain injury (Periventricular Leukomalacia (PVL) or Interventricular hemorrhage (IVH) on term corrected brain imaging prior to discharge in participants receiving additional caffeine compared to those receiving placebo.
Rates of Abnormal General Movement Assessment (GMA) | up to 6 months
  Rates of abnormal GMA prior to discharge in participants receiving additional caffeine compared to those receiving placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Harer, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will submit data to the National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH). NICHD DASH is a NICHD-funded controlled access data repository established to facilitate data sharing and access to biospecimens for all NICHD clinical research. This study will produce four data types: Clinical data, Urine proteomic biomarker, PK/PD data, and near infrared spectroscopy (NIRS) oxygenation data. The final clinical dataset will include demographic data and study-related tests obtained from the electronic medical record. The urine proteomic data will contain output from the biological urine samples from each research subject. The PK/PD data will contain caffeine serum concentration and renal oxygenation data at various timepoints, dose levels, and selected demographic and clinical data. The NIRS oxygenation dataset will include every 1 second kidney and cerebral oxygenation percentage generated/obtained from INVOS Medtronic NIRS 7100 devices.
Supporting Information: Study Protocol, SAP, ICF